CLINICAL TRIAL: NCT00847912
Title: CSP #562 - The VA Keratinocyte Carcinoma Chemoprevention Trial
Acronym: VAKCCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 562
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms; Skin Diseases; Neoplasms, Basal Cell; Neoplasms, Squamous Cell; Carcinoma
Keywords: NMSC; nonmelanoma skin cancer; topical 5-FU 5% cream; Neoplasms; Antineoplastic Agents; Therapeutic Uses; Dermatologic Agents; Neoplasms by Site; carcinoma, basal cell; carcinoma, squamous cell
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms; Skin Diseases; Neoplasms, Basal Cell; Neoplasms, Squamous Cell; Carcinoma; Neoplasms; Neoplasms by Site | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: 5-fluorouracil (Experimental): Group assigned to blinded 5-FU (5-fluorouracil) cream applied to face and ears twice daily for maximum of 56 doses
  Interventions: Drug: 5-fluorouracil
- Arm 2: Placebo (Placebo Comparator): Group assigned to blinded placebo, vehicle control cream applied to face and ears twice daily for maximum of 56 doses
  Interventions: Drug: Placebo, vehicle control

INTERVENTIONS:
Drug: 5-fluorouracil — Apply thin layer of topical 5-FU 5% cream twice daily to face and ears for 4 weeks. Treatment to be initiated immediately after randomization. If unable to tolerate the twice daily 5-FU, they will discontinue the treatment and initiate "cool-down" treatment with triamcinolone 0.1% cream twice daily until the symptoms resolve. At 3 weeks after stopping 5-FU, if and only if the participant has not received at least the minimum 2 week (28 dose) course, 5-FU treatment will be resumed on a once-daily basis to complete the 56 dose course. If this is not tolerated, the "cool-down" routine will be followed, but 5-FU will be stopped.
  Other Names: Efudex, 5-FU
  Arms: Arm 1: 5-fluorouracil
Drug: Placebo, vehicle control — Apply thin layer of vehicle control cream twice daily to face and ears for 4 weeks. Treatment to be initiated immediately after randomization. If unable to tolerate the twice daily vehicle control cream, they will discontinue the treatment and initiate "cool-down" treatment with triamcinolone 0.1% cream twice daily until the symptoms resolve. At 3 weeks after stopping vehicle control cream, if and only if the participant has not received at least the minimum 2 week (28 dose) course, vehicle control cream treatment will be resumed on a once-daily basis to complete the 56 dose course. If this is not tolerated, the "cool-down" routine will be followed, but vehicle control cream will be stopped.
  Other Names: Placebo
  Arms: Arm 2: Placebo

SUMMARY:
The main purpose of this study is to see if 5-fluorouracil (5-FU) skin cream can prevent the growth of new skin cancers on the face and ears. The cost of trying to prevent skin cancer will be compared to the usual cost of treating skin cancer. Participants are being asked to be a part of this study because the participants have been treated for two or more skin cancers within the past five (5) years. At least one of these cancers occurred on the face or ears. Having had two or more skins cancers in the past 5 years makes it likely that participants will develop additional skin cancers in the future.

Exposure to ultraviolet radiation from the sun or artificial sources such as tanning beds is a major cause of basal cell and squamous cell carcinoma of the skin. Using lotions, creams, or gels that contain sunscreens can help protect the skin from premature aging and damage that may lead to skin cancer.

The 5-FU skin cream used in this study is FDA-approved to treat some types of skin cancers and spots that might become skin cancer. However, 5-FU skin cream has never been studied to see if it can prevent skin cancer. This drug is not approved by the FDA for how it will be used in this study.

In this study, one half of the patients will use the 5-FU cream and the other half will use a skin cream that looks identical to the 5-FU cream but does not have 5-FU or any other active drug in it.

Approximately twelve VA medical centers will work together in this study. About one thousand (1000) patients will be in this study. The study is sponsored by the U.S. Department of Veterans Affairs Cooperative Studies Program.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) of the skin, both of which are keratinocyte carcinomas (KCs), account for a half of all cancers in the United States, and over 100,000 diagnoses per year in the VA. The standard treatment for these KCs is excision of the lesion, and they cost the US health care system some $2.5 billion annually and about $100 million annually in the VA. There is no proven means to prevent KCs (except perhaps for a modest benefit of intensive daily sunscreen use). An effective prevention strategy would dramatically change the way high-risk patients are managed and could substantially reduce the costs of care. The investigators' preliminary analysis indicates that the savings will be $116 per high-risk patient and will account for a total national savings of over $11 million. These findings imply that the study would pay for itself by the end of 4 years. The investigators hypothesize that topical 5-fluorouracil (5-FU) chemoprevention will prevent skin cancer surgeries and will be cost-saving. To test this the investigators propose a randomized controlled trial of 5-FU compared to a vehicle control to the face and ears in a high-risk population.

In the study, 1000 Veterans at high-risk of skin cancer defined as at least 2 KCs in the prior 5 years, at least one of which was on the face or ears, will be randomized to 5-FU or a vehicle control cream, and followed for 2 to 4 years. The primary endpoint will be surgery for any KC on the face and ears. The investigators will also assess the cost of care, quality of life, the side effects associated with treatment, and the prevalence and number of actinic keratoses, a skin cancer precursor and itself a cause of morbidity and cost. By targeting patients at high-risk, the study focuses on high-cost patients for whom this treatment could both improve outcomes (cancers and quality of life) and reduce costs.

ELIGIBILITY:
Inclusion Criteria:

* Veteran who is at high risk for developing skin cancer defined as 2 keratinocyte carcinomas in the past 5 years, at least one of which was located on the face or ears

Exclusion Criteria:

* Participants who are unable to speak English
* Participants with KC at randomization
* Participants currently using or having used field therapy for AKs on the face or ears in the past 3 years. The vast majority of these field treatments would have been with 5-FU cream. The investigators will allow recent use of therapies that are applied to individual AK lesions (e.g. cryotherapy), but not those that were used on an entire area (field) in the study treatment area Participants currently using or having used systemic 5-fluorouracil or oral capecitabine (Xeloda) within the past 3 years Participants with known allergy to sunscreen, triamcinolone and/or 5-fluorouracil.

Exclusions 6-l0: The investigators will exclude the small proportion who get their KCs for special reasons other than ultraviolet radiation exposure (see list below), since that etiologic difference, which is associated with a prognostic difference, could be associated with a biologic difference in response to chemoprevention efforts. These will include:

* Solid organ transplant recipients, such as renal, hepatic, or cardiac transplant patients
* Individuals with genetic disorders associated with very high cancer risk such as:
* basal cell nevus syndrome
* erythrodysplasia verruciformis
* xeroderma pigmentosum
* Arsenic exposure
* PUVA (Psoralen plus UVA) treatment
* Cutaneous T-cell lymphoma
* Prior or current radiation therapy to the face and/or ears.

Additional exclusions (12-15) are:

* Those who, in the opinion of the recruiting investigator, have very high mortality risk at randomization (less than 50% chance of surviving 4 years) due to co morbid illness such as metastatic cancer or COPD.
* For women of childbearing potential an initial pregnancy test and ongoing birth control will be required for participation.
* Patients with known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency by self report or noted in the medical record (they have increased toxicity from systemic 5-FU, although screening for this is not part of dermatologic practice and will not be part of this study).
* Patients on methotrexate (these will constitute about 1% of potentially eligible individuals) because they may have more severe reactions to topical 5-FU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2009-06-26 (Actual); Primary Completion 2013-06-28 (Actual); Study Completion 2016-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Weinstock, MD, Study Chair — Providence VA Medical Center, Providence, RI
Locations (13):
- United States (13):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KC, Lew R, Weinstock MA. Improvement in precision of counting actinic keratoses. Br J Dermatol. 2014 Jan;170(1):188-91. doi: 10.1111/bjd.12629. PMID 24102420
- [Background] Korgavkar K, Firoz EF, Xiong M, Lew R, Marcolivio K, Burnside N, Dyer R, Weinstock MA; VAKCC Trial Group. Measuring the severity of topical 5-fluorouracil toxicity. J Cutan Med Surg. 2014 Jul-Aug;18(4):229-35. doi: 10.2310/7750.2013.13143. PMID 25008439
- [Background] Pomerantz H, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin G, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri J, Lew R, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Long-term Efficacy of Topical Fluorouracil Cream, 5%, for Treating Actinic Keratosis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):952-60. doi: 10.1001/jamadermatol.2015.0502. PMID 25950503
- [Background] Chen SC, Hill ND, Veledar E, Swetter SM, Weinstock MA. Reliability of quantification measures of actinic keratosis. Br J Dermatol. 2013 Dec;169(6):1219-22. doi: 10.1111/bjd.12591. PMID 24033340
- [Result] Pomerantz H, Korgavkar K, Lee KC, Lew R, Weinstock MA; VAKCC Trial Group. Validation of Photograph-Based Toxicity Score for Topical 5-Fluorouracil Cream Application. J Cutan Med Surg. 2016 Sep;20(5):458-66. doi: 10.1177/1203475416643952. Epub 2016 Apr 18. PMID 27207349
- [Result] Siegel JA, Luber AJ, Weinstock MA; Department of Veterans Affairs Topical Tretinoin Chemoprevention Trial and Department of Veterans Affairs Keratinocyte Carcinoma Chemoprevention Trial Groups. Predictors of actinic keratosis count in patients with multiple keratinocyte carcinomas: A cross-sectional study. J Am Acad Dermatol. 2017 Feb;76(2):346-349. doi: 10.1016/j.jaad.2016.09.020. No abstract available. PMID 28088997
- [Result] Walker JL, Siegel JA, Sachar M, Pomerantz H, Chen SC, Swetter SM, Dellavalle RP, Stricklin GP, Qureshi AA, DiGiovanna JJ, Weinstock MA. 5-Fluorouracil for Actinic Keratosis Treatment and Chemoprevention: A Randomized Controlled Trial. J Invest Dermatol. 2017 Jun;137(6):1367-1370. doi: 10.1016/j.jid.2016.12.029. No abstract available. PMID 28532759
- [Result] Pomerantz H, Chren MM, Lew R, Weinstock MA; VA Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group*. Validation and comparison of quality-of-life measures for topical 5-fluorouracil treatment: results from a randomized controlled trial. Clin Exp Dermatol. 2017 Jul;42(5):488-495. doi: 10.1111/ced.13089. PMID 28621489
- [Result] Korgavkar K, Weinstock MA, Lee KC; VAKCC Trial Group. Evaluation of photoaging scales in an elderly male population. J Eur Acad Dermatol Venereol. 2017 Nov;31(11):e489-e490. doi: 10.1111/jdv.14330. Epub 2017 Jun 20. No abstract available. PMID 28500658
- [Result] Leader NF, Means AD, Robinson-Bostom L, Telang GH, Wilkel CS, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention Trial group. Interrater reliability for histopathologic diagnosis of keratinocyte carcinomas. J Am Acad Dermatol. 2018 Jan;78(1):185-187. doi: 10.1016/j.jaad.2017.07.024. No abstract available. PMID 29241779
- [Result] Korgavkar K, Lee KC, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Effect of Topical Fluorouracil Cream on Photodamage: Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2017 Nov 1;153(11):1142-1146. doi: 10.1001/jamadermatol.2017.2578. PMID 28877312
- [Result] Means AD, Lee KC, Korgavkar K, Swetter SM, Dellavalle RP, Chen S, Stricklin G, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Development of a Pigmented Facial Lesion Scale Based on Darkness and Extent of Lesions in Older Veterans. J Invest Dermatol. 2019 May;139(5):1185-1187. doi: 10.1016/j.jid.2018.11.017. Epub 2018 Nov 30. No abstract available. PMID 30508548
- [Result] Beatson M, Means AD, Leader NF, Robinson-Bostom L, Weinstock MA. Characteristics of Keratinocyte Carcinomas and Patients with Keratinocyte Carcinomas Following a Single 2-4 Week Course of Topical 5-fluorouracil on the Face and Ears. Acta Derm Venereol. 2019 Jun 1;99(7):707-708. doi: 10.2340/00015555-3176. No abstract available. PMID 30896781
- [Result] Beatson M, Siegel JA, Chren MM, Weinstock MA. Effects of increased actinic keratosis count on skin-related quality of life: results from the Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial. Eur J Dermatol. 2019 Oct 1;29(5):507-510. doi: 10.1684/ejd.2019.3637. PMID 31647464
- [Result] Beatson M, Misitzis A, Landow S, Yoon J, Higgins HW 2nd, Phibbs C, Weinstock MA. Predictors of Basal Cell Carcinoma and Implications for Follow-Up in High-Risk Patients in the Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial. J Cutan Med Surg. 2021 Jan-Feb;25(1):102-103. doi: 10.1177/1203475420945230. Epub 2020 Sep 3. No abstract available. PMID 32880186
- [Result] Misitzis A, Stratigos AJ, Beatson M, Mastorakos G, Dellavalle RP, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention Trial Group. The association of metformin use with keratinocyte carcinoma development in high-risk patients. Dermatol Ther. 2020 Nov;33(6):e14402. doi: 10.1111/dth.14402. Epub 2020 Oct 20. PMID 33047438
- [Result] Siegel JA, Chren MM, Weinstock MA; Department of Veterans Affairs Keratinocyte Carcinoma Chemoprevention Trial Group. Correlates of skin-related quality of life (QoL) in those with multiple keratinocyte carcinomas (KCs): A cross-sectional study. J Am Acad Dermatol. 2016 Sep;75(3):639-642. doi: 10.1016/j.jaad.2016.05.008. No abstract available. PMID 27543222
- [Result] Yoon J, Phibbs CS, Chow A, Pomerantz H, Weinstock MA. Costs of Keratinocyte Carcinoma (Nonmelanoma Skin Cancer) and Actinic Keratosis Treatment in the Veterans Health Administration. Dermatol Surg. 2016 Sep;42(9):1041-7. doi: 10.1097/DSS.0000000000000820. PMID 27465252
- [Derived] Weinstock MA, Thwin SS, Siegel JA, Marcolivio K, Means AD, Leader NF, Shaw FM, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin GP, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri JE, Robinson-Bostom L, Ringer RJ, Lew RA, Ferguson R, DiGiovanna JJ, Huang GD; Veterans Affairs Keratinocyte Carcinoma Chemoprevention Trial (VAKCC) Group. Chemoprevention of Basal and Squamous Cell Carcinoma With a Single Course of Fluorouracil, 5%, Cream: A Randomized Clinical Trial. JAMA Dermatol. 2018 Feb 1;154(2):167-174. doi: 10.1001/jamadermatol.2017.3631. PMID 29299592

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Placebo, Vehicle Control: Group assigned to blinded placebo, vehicle control cream applied to face and ears twice daily for maximum of 56 doses
  Placebo, vehicle control: Apply thin layer of vehicle control cream twice daily to face and ears for 4 weeks. Treatment to be initiated immediately after randomization. If unable to tolerate the twice daily vehicle control cream, they will discontinue the treatment and initiate "cool-down" treatment with triamcinolone 0.1% cream twice daily until the symptoms resolve. At 3 weeks after stopping vehicle control cream, if and only if the participant has not received at least the minimum 2 week (28 dose) course, vehicle control cream treatment will be resumed on a once-daily basis to complete the 56 dose course. If this is not tolerated, the "cool-down" routine will be followed, but vehicle control cream will be stopped.
Period: Overall Study
Arm/Group | Arm 1: 5-fluorouracil | Arm 2: Placebo, Vehicle Control
Started | 477 | 477
Completed | 468 | 464
Not Completed | 9 | 13
Not completed — Protocol Violation | 6 | 7
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 5-fluorouracil | Arm 2: Placebo, Vehicle Control | Total
Number analyzed (Participants) | 468 | 464 | 932
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (9.2) | 71.5 (9.4) | 71.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 457 | 459 | 916
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 464 | 459 | 923
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 455 | 457 | 912
  More than one race | 10 | 4 | 14
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 468 | 464 | 932

OUTCOME MEASURES:

1. Primary Outcome: The Time to Diagnosis of the First Keratinocyte Carcinoma (KC) on the Face or Ears for Which Surgery is Performed
Description: Diagnosis of the first Primary Basil Cell Carcinoma (BCC) or primary Squamous Cell Carcinoma (SCC) on the face or ears that was removed surgically.
Time Frame: From randomization to last visit prior to end of study date (6/30/2013), assessed up to four years
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Arm 1: 5-fluorouracil: Group assigned to blinded 5-fluorouracil (5-FU) cream applied to face and ears twice daily for maximum of 56 doses
  5-fluorouracil: Apply thin layer of topical 5-FU 5% cream twice daily to face and ears for 4 weeks. Treatment to be initiated immediately after randomization. If unable to tolerate the twice daily 5-FU, they will discontinue the treatment and initiate "cool-down" treatment with triamcinolone 0.1% cream twice daily until the symptoms resolve. At 3 weeks after stopping 5-FU, if and only if the participant has not received at least the minimum 2 week (28 dose) course, 5-FU treatment will be resumed on a once-daily basis to complete the 56 dose course. If this is not tolerated, the "cool-down" routine will be followed, but 5-FU will be stopped.
Arm/Group | Arm 1: 5-fluorouracil | Arm 2: Placebo, Vehicle Control
Number analyzed (Participants) | 468 | 464
years | 3.37 [3.21 to NA] — Upper 95% confidence interval could not be estimated due to an insufficient number of participants with events | 3.52 [3.08 to 3.70]
Statistical Analysis 1: Comparison: Arm 1: 5-fluorouracil vs Arm 2: Placebo, Vehicle Control; Test type: Superiority or Other; p = 0.93, Log Rank

2. Primary Outcome: Hazard Ratio for Surgically Treated KC
Time Frame: date of randomization to last visit before end of study follow up (6/30/2013), assessed up to four years
Measure: Number; unit: participants
Arm/Group | Arm 1: 5-fluorouracil | Arm 2: Placebo, Vehicle Control
Number analyzed (Participants) | 468 | 464
participants | 182 | 177
Statistical Analysis 1: Comparison: Arm 1: 5-fluorouracil vs Arm 2: Placebo, Vehicle Control; Test type: Superiority or Other; p = 0.93, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.82 to 1.24]

ADVERSE EVENTS:
Time Frame: Active monitoring of Adverse Events and Serious Adverse Events began when the participant signed the Consent Form. Adverse Event data collection ended when the participant ended study participation, and Serious Adverse Event data collection continued until 30 days after study participation ended, assessed up to four years.
Description: Adverse events collected were those related to the study intervention. Data on adverse events were collected spontaneously through patient reports, actively elicited at each clinic visit through open ended questionings and examination, and gathered at the time of telephone contact during the therapy period. All serious adverse events were collected, including those considered related and unrelated to the study interventions.Subjects were monitored for SAE at each study visit and telephone call.
Arm/Group | Arm 1: 5-fluorouracil | Arm 2: Placebo
Serious Adverse Events (participants affected / at risk) | 190/468 | 190/464
Other Adverse Events (participants affected / at risk) | 451/468 | 227/464
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 5-fluorouracil (N=468) | Arm 2: Placebo (N=464)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 5 (5)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2)
Angina unstable (Cardiac disorders) | 5 (5) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 13 (16)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (2)
Bradycardia (Cardiac disorders) | 2 (3) | 3 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 7 (11) | 7 (8)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 5 (6) | 14 (17)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 7 (7)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (3)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adhesion (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 8 (10) | 10 (10)
Death (General disorders) | 4 (4) | 6 (6)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (4) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 4 (6)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis (Infections and infestations) | 1 (2) | 0 (0)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (20) | 21 (26)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (13) | 8 (9)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Cardiac monitoring (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (12) | 11 (11)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 5 (6)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (5)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1)
Basilar artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 7 (7)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 2 (4)
Dementia (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Moyamoya disease (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Adjustment disorder with anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Binge drinking (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (3) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (4)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 4 (6)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 9 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respite care (Social circumstances) | 0 (0) | 1 (2)
Social stay hospitalisation (Social circumstances) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 2 (2)
Elective procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device change (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Parotidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Plasmapheresis (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Skin graft (Surgical and medical procedures) | 1 (1) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Vena cava filter insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 5 (5)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 5-fluorouracil (N=468) | Arm 2: Placebo (N=464)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 3 (3) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 4 (4) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Iris cyst (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 11 (12) | 6 (6)
Pyrexia (General disorders) | 1 (1) | 1 (2)
Swelling (General disorders) | 0 (0) | 3 (3)
Syringe issue (General disorders) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0)
Tenderness (General disorders) | 2 (2) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (5) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 4 (4)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Emergency care examination (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tunnel vision (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 22 (25) | 2 (2)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 447 (495) | 187 (218)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Oral surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 7 (7) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes